CLINICAL TRIAL: NCT01690312
Title: Clinical Study to Assess the Acute and Chronic Effects of a High-DHA Fish Oil on Fasting and Post-Prandial Biomarkers of Cardiovascular Disease Risk in Adults on Statin Therapy.
Brief Title: Clinical Study to Assess High-DHA Fish Oil on Biomarkers of Cardiovascular Disease Risk in Adults on Statin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Collaborators: Biodroga Inc. (Industry); University of Guelph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-09-002; 150038 (Other: Health Canada)
Record Dates: First submitted 2012-09-10; First posted 2012-09-21 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Disease
Keywords: Humans; Cardiovascular Disease; Statins; Fish Oil; DHA; EPA; High-DHA; Triglycerides; Total cholesterol [TC]; Lipoproteins; High-density lipoprotein [HDL2, HDL3]; Low-density lipoprotein [LDL1+2+3+4]; Lipoprotein A [Lp(a)]; Intermediate-density lipoprotein (IDL); Very low-density lipoprotein (VLDL1+2, VLDL3); Remnant Lipoproteins; High-sensitivity C-Reactive Protein [hs-CRP]; Homocysteine; Essential Fatty Acid Profile; Apolipoprotein B; Apolipoprotein A-1; Glucose; Insulin; Fasted; Post-Prandial
MeSH Terms: conditions — Cardiovascular Diseases; Huntington Disease-Like 2; Insulin Resistance | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Dietary Supplement - Fish Oil) (Experimental): On Day 1 & Day 29, the researcher will obtain anthropometric measurements as specified in the study protocol. A venous catheter will be inserted and a fasted blood sample will be drawn, which will be analyzed for study primary and secondary endpoints. Participants will consume a Breakfast Meal (which will represent t0) and will have blood drawn at a total of 7 time points. Blood samples drawn at30, t60, t120, and t180 will be analyzed for glucose and insulin; blood samples drawn at t60, t120, t180, t240, t300 and t360 will be analyzed for triglycerides. Upon completion of the 6 hour blood draw period, the venous catheter will be removed.
  On Day 15, the researcher will obtain anthropometric measurements as specified in the study protocol.
  Interventions: Dietary Supplement: Fish Oil
- 2 (Placebo) (Experimental): On Day 1 & Day 29, the researcher will obtain anthropometric measurements as specified in the study protocol. A venous catheter will be inserted and a fasted blood sample will be drawn, which will be analyzed for study primary and secondary endpoints. Participants will consume a Breakfast Meal (which will represent t0) and will have blood drawn at a total of 7 time points. Blood samples drawn at30, t60, t120, and t180 will be analyzed for glucose and insulin; blood samples drawn at t60, t120, t180, t240, t300 and t360 will be analyzed for triglycerides. Upon completion of the 6 hour blood draw period, the venous catheter will be removed.
  On Day 15, the researcher will obtain anthropometric measurements as specified in the study protocol.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — On Day 1 and Day 15, participants will receive a 2-week supply of study supplements and will be instructed to consume 4 capsules per day. Each capsule contains 1000 mg of fish oil [620 mg of DHA and 150 mg of EPA], providing a total daily dosage of 4000 mg of fish oil [3080 mg of DHA+EPA].
  Arms: 1 (Dietary Supplement - Fish Oil)
Dietary Supplement: Placebo — On Day 1 and Day 15, participants will receive a 2-week supply of study supplements and will be instructed to consume 4 capsules per day. Each capsule contains 1000 mg of olive oil, providing a total daily dosage of 4000 mg of olive oil.
  Arms: 2 (Placebo)

SUMMARY:
The objective of this study is to determine the acute and chronic [4-week] effects of a high-DHA fish oil supplement on fasting and post-prandial (post-meal) biomarkers of cardiovascular disease risk, in adults on Statin therapy.

DETAILED DESCRIPTION:
This study involves fasted and post-prandial components.

Fasted Study:

Participants will provide fasting blood samples pre-and post-intervention [4-week administration of supplement or placebo] in Treatment Period I. Participants will again provide fasting blood samples pre-and post-intervention [4-week administration of supplement or placebo, opposite to Treatment Period I] during Treatment Period II.

There will be a 4-week washout period during the two Treatment Periods.

Post-prandial study:

Participants will also complete a post-prandial study pre-and post-intervention during each Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult between the ages of 18 and 70;
* Be a male or a post-menopausal female who has gone a minimum of one year since their last menses;
* Be taking Statin medication at a stable dose for a minimum of four weeks prior to study commencement [and whom have reached a target LDL level];
* Have elevated fasting triglyceride levels [greater than 1.5 mmol/L but less than 5.7 mmol/L];
* Have fasting blood glucose levels below the study cut-off [less than 7.0 mmol/L];
* Have a Body Mass Index (BMI) less than 35.0
* Be taking natural health products BUT agree to cease consumption during the study period and a 4-week pre-study washout prior to study commencement. Study participants will be allowed to consume a daily multivitamin if they have been doing so at a stable dose for a minimum of three months prior to study commencement.

Exclusion Criteria:

* Be younger than 18 years of age or older than 70 years of age;
* Be an adult pre- or peri-menopausal female;
* Not have taken Statin medication at a stable dose for a minimum of 4 weeks prior to study commencement;
* Have fasting triglyceride levels outside of study limits[ie/ less than 1.5 mmol/L or greater than 5.7 mmol/L];
* Have elevated fasting blood glucose levels [greater or equal to 7.0 mmol/L];
* Have high blood pressure [greater than 140/100]
* Have a Body Mass Index (BMI) equal to or greater than 35.0
* Have a pre-existing cardiovascular disease or illness, including angina, myocardial infarction, stroke, intermittent claudication or transient ischemic attack;
* Have a known allergy to fish and/or fish oil, olive oil, soy or Vitamin E;
* Be taking natural health products but are unwilling to cease consumption during the study period and a 4-week pre-study washout prior to study commencement;
* Consume more than two (2) fish meals on a weekly basis
* Consume excessive amounts of alcohol on a weekly basis [more than 10 alcoholic drinks per week];
* Anticipate or have planned surgery during the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Triglyceride [TG] | 0 and 4 weeks
  Fasted and postprandial samples will be drawn (hourly up to 6 hours).

SECONDARY OUTCOMES:
Glucose | 0 and 4 weeks
  Fasted and postprandial samples will be drawn (every 30 minutes up to 2 hours).
Insulin | 0 and 4 weeks
  Fasted and postprandial samples will be drawn (every 30 minutes up to 2 hours).
Total cholesterol [TC] | 0 and 4 weeks
  A fasted blood sample will be taken.
High-density lipoprotein [HDL] | 0 and 4 weeks
  A fasted blood sample will be taken.
Low-density lipoprotein [LDL] | 0 and 4 weeks
  A fasted blood sample will be taken.
Very low-density lipoprotein [VLDL] | 0 and 4 weeks
  A fasted blood sample will be taken.
Lipoprotein A | 0 and 4 weeks
  A fasted blood sample will be taken.
Intermediate-density lipoprotein [IDL] | 0 and 4 weeks
  A fasted blood sample will be taken.
Remnant Lipoproteins | 0 and 4 weeks
  A fasted blood sample will be taken.
High-sensitivity C-Reactive Protein [hs-CRP] | 0 and 4 weeks
  A fasted blood sample will be taken.
Homocysteine | 0 and 4 weeks
  A fasted blood sample will be taken.
Essential Fatty Acid Profile | 0 and 4 weeks
  A fasted blood sample will be taken.
Apolipoprotein B | 0 and 4 weeks
  A fasted blood sample will be taken.
Apolipoprotein A-1 | 0 and 4 weeks
  A fasted blood sample will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Duncan, Ph.D., R.D., Principal Investigator — University of Guelph
Locations (1):
- Nutrasource Diagnostics Inc., Guelph, Ontario, Canada